CLINICAL TRIAL: NCT02843828
Title: Gait Pattern Analysis and Feasibility of Gait Training With a Newly Developed Walking Assist Robot in Stroke Patients and Elderly Adults
Brief Title: Gait Pattern Analysis and Feasibility of Gait Training With a Walking Assist Robot in Stroke Patients and Elderly Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Collaborators: Samsung Electronics (Industry)
Responsible Party: Principal Investigator, Yun-Hee Kim, Professor, MD, PhD, Samsung Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2015-05-013-003
Record Dates: First submitted 2016-07-14; First posted 2016-07-26 (Estimated); Last update posted 2019-04-10 (Actual); Status verified 2019-04

CONDITIONS: Stroke; Healthy
Keywords: Exoskeleton Device; elderly; stroke; gait rehabilitation
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Samsung Hip Assist v1 (Experimental): gait rehabilitation with Samsung Hip Assist v1 10 sessions (5sessions - treadmill gait training / 5sessions - overground gait training), 30 min per session
  Interventions: Device: gait rehabilitation with Samsung Hip Assist v1
- Conventional gait training (Active Comparator): gait rehabilitation without Samsung Hip Assist v1 10 sessions (5sessions - treadmill gait training / 5sessions - overground gait training), 30 min per session
  Interventions: Other: gait rehabilitation without Samsung Hip Assist v1

INTERVENTIONS:
Device: gait rehabilitation with Samsung Hip Assist v1 — Participants will participate in 10 sessions of gait rehabilitation with Samsung Hip Assist v1 (5sessions-treadmill gait training / 5sessions-overground gait training), 30min per session
  Arms: Samsung Hip Assist v1
Other: gait rehabilitation without Samsung Hip Assist v1 — Participants will participate in 10 sessions of gait rehabilitation without Samsung Hip Assist v1 (5sessions-treadmill gait training / 5sessions-overground gait training), 30min per session
  Arms: Conventional gait training

SUMMARY:
The purpose of this study was to investigate the effects of the new wearable hip assist robot developed by Samsung Advanced Institute of Technology (Samsung Electronics Co, Ltd., Korea) to gait rehabilitation in elderly adults and stroke patients.

DETAILED DESCRIPTION:
Randomized, two treatment groups

Number of Subjects : 54 subjects (n=27 per group)

Group 1 : gait rehabilitation with hip assist robot / 10 sessions (5sessions - treadmill gait training / 5sessions - overground gait training), 30min per session

Group 2 : gait rehabilitation without hip assist robot / 10 sessions (5sessions - treadmill gait training / 5sessions - overground gait training), 30min per session

Primary objective is to demonstrate the effects of hip assist robot on spatio-temporal parameters measured by motion capture system (Motion Analysis Corporation, Santa Rosa, CA, USA), muscle activation patterns measured by surface electromyography (sEMG) (Noraxon Inc., Scottsdale, AZ, USA), metabolic energy cost parameters measured by portable cardiopulmonary metabolic system (Cosmed K4B2, Rome, Italy) and foot pressure distribution measured by F-Scan Mobile system (Tekscan Inc., South Boston, MA, USA).

Secondary objective is to demonstrate the effects of hip assist robot on motor function improvement evaluated by Berg Balance Scale (BBS), Tinetti performance oriented mobility assessment (POMA), Korean version Modified Bathel index (K-MBI), Modified Rankin Scale (MRS), Functional Ambulation Classification (FAC), Fugl-Meyer assessment for lower extremity (FMA), Korean version Fall Efficacy Scale (K-FES), Manual Muscle Test (MMT) and Range of Motion (ROM).

ELIGIBILITY:
Inclusion Criteria:

* Elderly adults

  1. Age: between 65 and 84 years
  2. elderly adults who had no neurological or musculoskeletal abnormalities affecting gait
  3. Ability to walk at least 10m regardless of assist devices
  4. High levels of physical performance (SPPB > 7)
  5. Subject is willing to be randomized to the control group or the treatment group
* Stroke

  1. Age: between 50 and 84 years
  2. ≥ 3 months post stroke
  3. Ability to walk at least 10m regardless of assist devices
  4. Adequate gait function (FAC > 3)
  5. Physician approval for patient participation
  6. Subject is willing to be randomized to the control group or the treatment group

Exclusion Criteria:

* Elderly adults

  1. History of any diseases (eg. lower extremity orthopedic diseases, neurologic disorders, cardiovascular disease, heart failure, uncontrolled hypertension that affect walking capacity, efficiency, and endurance)
  2. Severe visual impairment or dizziness that increases the risk of falls
* Stroke

  1. Serious cardiac conditions (hospitalization for myocardial infarction or heart surgery within 3 months, history of congestive heart failure, documented serious and unstable cardiac arrhythmias, hypertrophic cardiomyopathy, severe aortic stenosis, angina or dyspnea at rest or during activities of daily living)
  2. Advanced liver, kidney, cardiac, or pulmonary disease
  3. History of concussion in last 6 months
  4. History of unexplained, recurring headaches, epilepsy/seizures/skull fractures or skull deficits
  5. Preexisting neurological disorders such as Parkinson's disease, Amyotrophic Lateral Sclerosis (ALS), Multiple Sclerosis (MS), dementia

Ages: 50 Years to 84 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2016-01-02 (Actual); Primary Completion 2017-08-30 (Actual); Study Completion 2017-09-01 (Actual)

PRIMARY OUTCOMES:
Change in 10 meter walk test from baseline in gait speed | session 0 (initial visit); session 11 (at approximately 4 weeks)
  Measure of self selected speeds by measuring the time it takes an individual to walk 10 meters. To perform the test, patient walks 10 meters (33 ft) and the time is measured when the leading foot crosses the start line and the finish line. The instructions are: "Please walk this distance at your normal pace when I say go."

SECONDARY OUTCOMES:
Berg Balance Scale (BBS) | session 0 (initial visit); session 11 (at approximately 4 weeks)
  The BBS is a 14-item objective measure designed to assess static balance and fall risk in adult populations and is a well-accepted measure in the stroke literature. The functional activities that are assessed include sitting and standing balance during transfers, altered base of support, reaching, turning, eyes open and closed.
Tinetti performance oriented mobility assessment (POMA) | session 0 (initial visit); session 11 (at approximately 4 weeks)
  Task-oriented outcome measure that assesses gait and balance ability is composed of a 9-item gait portion (POMA-G) and 7-item balance portion (POMA-B).
Modified Bathel index (MBI) | session 0 (initial visit); session 11 (at approximately 4 weeks)
  The MBI is a measure of activities of daily living, which shows the degree of independence of a patient from any assistance. It covers 10 domains of functioning (activities): bowel control, bladder control, as well as help with grooming, toilet use, feeding, transfers, walking, dressing, climbing stairs, and bathing.
Modified Rankin Scale (MRS) | session 0 (initial visit); session 11 (at approximately 4 weeks)
  The modified Rankin Scale (mRS) is a commonly used scale for measuring the degree of disability or dependence in the daily activities of people who have suffered a stroke or other causes of neurological disability.
Functional Ambulation Classification (FAC) | session 0 (initial visit); session 11 (at approximately 4 weeks)
  The Functional Ambulation Categories (FAC) is a functional walking test that evaluates ambulation ability. This 6-point scale assesses ambulation status by determining how much human support the patient requires when walking, regardless of whether or not they use a personal assistive device.
Fugl-Meyer assessment for lower extremity (FMA) | session 0 (initial visit); session 11 (at approximately 4 weeks)
  The Fugl-Meyer Assessment (FMA) is a stroke-specific, performance-based impairment index. It is designed to assess motor functioning, balance, sensation and joint functioning in patients with post-stroke hemiplegia. It is applied clinically and in research to determine disease severity, describe motor recovery, and to plan and assess treatment.
Fall Efficacy Scale (FES) | session 0 (initial visit); session 11 (at approximately 4 weeks)
  Fall Efficacy Scale (FES) is a 10-item questionnaire designed confidence in their ability to perform 10 daily tasks without falling as an indicator of how one's fear of falling impacts physical performance. Each item is rated from 1 ("very confident") to 10 ("not confident at all"), and the per item ratings are added to generate a summary total score.
Manual Muscle Test (MMT) | session 0 (initial visit); session 11 (at approximately 4 weeks)
  Manual muscle testing (MMT) is a procedure for the evaluation of the function and strength of individual muscles and muscle groups based on the effective performance of a movement in relation to the forces of gravity and manual resistance.
Range of Motion (ROM) | session 0 (initial visit); session 11 (at approximately 4 weeks)
  Range of Motion (ROM) testing is the measurement of movement around a specific joint or body part.

CONTACTS AND LOCATIONS:
Overall Officials: Yun-Hee Kim, MD, PhD, Study Chair — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lee HJ, Lee SH, Seo K, Lee M, Chang WH, Choi BO, Ryu GH, Kim YH. Training for Walking Efficiency With a Wearable Hip-Assist Robot in Patients With Stroke: A Pilot Randomized Controlled Trial. Stroke. 2019 Dec;50(12):3545-3552. doi: 10.1161/STROKEAHA.119.025950. Epub 2019 Oct 18. PMID 31623545
- [Derived] Lee SH, Lee HJ, Chang WH, Choi BO, Lee J, Kim J, Ryu GH, Kim YH. Gait performance and foot pressure distribution during wearable robot-assisted gait in elderly adults. J Neuroeng Rehabil. 2017 Nov 28;14(1):123. doi: 10.1186/s12984-017-0333-z. PMID 29183379